CLINICAL TRIAL: NCT02071550
Title: 10cmH2O Peep Application and Cerebral Oxygenation in Laparoscopic Surgery: a Comparative Study With Invos and Foresight Devices
Acronym: NIRS AND PEEP
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, aslı demir, Associated professor, Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 10869
Record Dates: First submitted 2014-02-18; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: laparoscopic cholecystectomy, near infrared spectroscopy, positive end expiratory pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- zero PEEP: Patients undergoing laparoscopic cholecystectomy and monitorized with FORESIGHT,INVOS monitor
  Interventions: Device: FORESİGHT cerebral oxygen monitor and INVOS cerebral oxygen monitor; Device: FORESIGHT and INVOS monitor
- 10 CM H2O PEEP: Patients undergoing laparoscopic cholecystectomy and monitorized with FORESIGHT,INVOS monitor
  Interventions: Device: FORESİGHT cerebral oxygen monitor and INVOS cerebral oxygen monitor; Device: FORESIGHT and INVOS monitor

INTERVENTIONS:
Device: FORESİGHT cerebral oxygen monitor and INVOS cerebral oxygen monitor
Device: FORESIGHT and INVOS monitor

SUMMARY:
In this study the investigators investigated changes in hemodynamic parameters and cerebral oxygen saturation (rSO2) associated with 10 cmH2O PEEP, which is assumed beneficial for the respiratory functions and oxygenation during the laparoscopic cholecystectomy (LC) applied at the 30°head-up left side position, is compared with using two individual devices (INVOS-FORESIGHT).

Methods: Afterwards the ethics committee approval of the hospital and receiving the written patients' consents, patients to undergo ASA I-II group elective laparoscopic surgery were randomly divided into two groups. Sensors of INVOS and FORESIGHT devices were placed on the right side forehead region. Totally 11 evaluation periods were formed, respectively: Pre-induction (1st Period), post-induction (2nd period), abdominal insufflation outset (3rd period): post-insufflation 5-minute intervals (4th, 5th, 6th, 7th 8th period), end of insufflation (9th period), end of operation (10th period) and end of anaesthesia (11th period). While one of the groups was not applied PEEP(ZEEP), the other group was applied 10 cmH2O simultaneously with the abdominal insufflation proceeding. Demographic data, hemodynamic values and rSO2 values were recorded for both groups at all 11 periods.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologist) class I and II
* Patients undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* ASA class III and IV
* Morbid obesity
* Emergency cases
* Cases returned to laparotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in cerebral oxymetry during laparoscopy | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey Yuksek Ihtisas Education and Research Hospital, Anesthesiology Clinic, Ankara, Turkey (Türkiye)